CLINICAL TRIAL: NCT07066254
Title: A Randomized Controlled Trial on the Effect of a Silver-impregnated Antimicrobial Foam Dressing on Surgical Site Infections After Cesarean Delivery
Brief Title: The Mepilex Cesarean Delivery Trial
Acronym: MEPIDEL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-16900
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Surgical Site Infection Following Cesarean Delivery
Keywords: Surgical site infection; Surgical Wound Infection; Postoperative Complications; Cesarean Section; Obstetric Surgical Procedures; Pregnant Women; Wound Dressing; Randomized Controlled Trial; Patient satisfaction; Anti-Infective Agents, Local; Infection Control; silver antimicrobial foam; mepilex
MeSH Terms: conditions — Surgical Wound Infection; Postoperative Complications; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized in a 1:1 ratio to receive either Mepilex Ag or the standard surgical dressing post-cesarean delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Surgical Dressing (Telfa non-adhesive pad, gauze, Primapore adhesive bandage) (Active Comparator): Participants in this arm will receive the standard postoperative surgical dressing currently used at our institution following cesarean delivery. This dressing consists of a Telfa non-adhesive pad placed over the incision, covered with gauze, and secured with a Primapore adhesive bandage.
  Interventions: Device: Standard Surgical Dressing (Telfa non-adhesive dressing, gauze, and Primapore adhesive bandage)
- Mepilex Ag Dressing (Experimental): Participants in this arm will receive a silver-impregnated antimicrobial foam dressing (Mepilex Ag) applied to the surgical incision following cesarean delivery.
  Interventions: Device: Mepilex Ag Dressing

INTERVENTIONS:
Device: Mepilex Ag Dressing — A silver-impregnated antimicrobial foam dressing (Mepilex Ag) will be placed over the cesarean incision immediately following skin closure in the operating room. Participants assigned to this intervention will be instructed to leave the dressing in place for 7 days, in accordance with manufacturer guidelines, unless earlier removal is necessary due to dressing saturation, displacement, or clinical concern. Mepilex Ag is FDA-cleared for use as a wound dressing and is designed to maintain a moist wound environment while providing sustained antimicrobial protection to help reduce the risk of surgical site infection.
  Other Names: Mepilex; Mepilex Ag; silver-impregnated antimicrobial foam
  Arms: Mepilex Ag Dressing
Device: Standard Surgical Dressing (Telfa non-adhesive dressing, gauze, and Primapore adhesive bandage) — A standard postoperative dressing consisting of a sterile Telfa non-adhesive pad placed over the cesarean incision, covered with gauze, and secured with a Primapore adhesive bandage. The dressing is applied immediately following skin closure in the operating room as part of routine institutional care. It is typically removed within 24 to 48 hours postoperatively, depending on wound condition and provider discretion.
  Other Names: Telfa; Primapore; adhesive bandage; standard dressing; unmedicated dressing
  Arms: Standard Surgical Dressing (Telfa non-adhesive pad, gauze, Primapore adhesive bandage)

SUMMARY:
The goal of this clinical trial is to learn whether using a silver-containing antimicrobial foam dressing (Mepilex Ag) can help prevent surgical site infections in patients undergoing cesarean delivery. The main questions it aims to answer are:

1. Does Mepilex Ag reduce the rate of surgical site infections after cesarean delivery?
2. Is Mepilex Ag more effective than standard wound dressings in preventing infection?

Researchers will compare those who receive the Mepilex Ag dressing to those who receive the standard dressing to see if the silver impregnated antimicrobial foam dressing lowers infection rate.

Participants will:

1. Undergo a routine cesarean delivery as per usual obstetric indication
2. Be randomly assigned to receive either a silver-containing foam dressing or a standard dressing after surgery
3. Be monitored for wound complications and signs of infection during the postpartum period

DETAILED DESCRIPTION:
Surgical site infections (SSIs) are among the most common complication following cesarean delivery and are associated with increased maternal morbidity, prolonged hospital stays, and higher healthcare costs. Despite the use of prophylactic antibiotics and standard perioperative practices, the risk of postoperative wound infection remains significant, especially in patients with additional risk factors such as obesity or diabetes.

Mepilex Ag is a silver-impregnated antimicrobial foam dressing that has antimicrobial properties and has been shown in other surgical populations to reduce the incidence of SSIs. It is FDA-cleared for use as a wound dressing but has not been specifically studied in the obstetrics population.

The overarching aim of this study is to assess whether the application of a silver-impregnated antimicrobial foam dressing at the time of cesarean delivery reduces the incidence of postoperative wound infections and improves related outcomes compared to standard surgical dressings. This randomized controlled trial will enroll eligible pregnant individuals undergoing cesarean delivery and randomly assign them to receive either the silver dressing or standard care dressing.

Study procedures and follow-up have been designed to systematically capture data related to postoperative wound outcomes, healthcare utilization, and patient experience. These data will support evaluation of the primary and secondary objectives and inform clinical practice regarding optimal strategies for wound management in this population.

This study aims to provide evidence to guide postoperative wound management after cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Undergoing non-emergent cesarean delivery at Montefiore-Einstein
* Able to provide informed consent in English or Spanish
* Has a working telephone number for follow-up communication

Exclusion Criteria:

* Known hypersensitivity or allergy to silver, Mepilex Ag, or adhesive materials
* Presence of active skin infection or open skin condition at the planned dressing site
* Psoriasis, eczema, or other acute or chronic dermatitis or skin condition that might affect the choice of optimal dressing or the results of the study
* Participation in another interventional trial affecting wound healing or surgical outcomes
* Immunocompromised status (e.g., current chemotherapy, chronic steroid use, or known HIV with CD4 <200)
* Intraoperative conversion to vertical skin incision or other nonstandard approach
* Inability to complete follow-up due to anticipated relocation, incarceration, or other logistical barrier

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Surgical Site Infection (SSI) Within 30 Days Post-Cesarean Delivery | Within 30 days of cesarean delivery/wound dressing application
  The primary outcome is the occurrence of a surgical site infection (SSI) within 30 days following cesarean delivery, as defined by the Centers for Disease Control and Prevention (CDC) criteria. Occurrences of SSIs include superficial incisional, deep incisional, or organ/space infections related to the surgical incision. Diagnosis will be determined through inpatient clinical monitoring, review of electronic health records for any related outpatient or emergency department visits, and follow-up telephone assessment conducted 30 days after cesarean delivery. SSIs will be summarized by study arm using descriptive statistics.

SECONDARY OUTCOMES:
Patient Satisfaction With Postoperative Dressing | At time of dressing removal, up to 7 days after cesarean delivery
  Patient satisfaction will be assessed using the Adapted Wound Dressing Satisfaction Questionnaire (WDSQ), a 9-item instrument that evaluates comfort, ease of movement, perceived wound protection, dressing appearance, and skin irritation. Responses to the first 8 questions are rated on a 5-point Likert scale, ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). The final item is rated on an 11-point Likert scale, ranging from 0 (Not at all satisfied) to 10 (Extremely satisfied), for an overall possible scoring range of 8-50, wherein higher scores are associated with increased global satisfaction with the assigned dressing.
Occurrence of Wound Seroma Formation | Within 30 days of cesarean delivery/wound dressing application
  Presence of a wound seroma at the surgical site, identified through documentation in the medical record within the 30 day postoperative period, will be summarized by study arm using basic descriptive statistics.
Occurrence of Wound Hematoma Formation | Within 30 days of cesarean delivery/wound dressing application
  Presence of a wound hematoma at the surgical site, identified through documentation in the medical record within the 30-day postoperative period, will be summarized by study arm using basic descriptive statistics.
Occurrence of Wound Dehiscence | Within 30 days of cesarean delivery/wound dressing application
  Presence of partial or complete wound dehiscence at the surgical site, identified through documentation in the medical record within the 30-day postoperative period, will be summarized by study arm using basic descriptive statistics.
Unscheduled Postoperative Healthcare Visits Related to Wound Concerns | Within 30 days of cesarean delivery/wound dressing application
  The number of unscheduled patient visits (either emergency department or outpatient clinic) related to wound complications, including concerns about drainage, infection, dehiscence, or dressing problems will be summarized by study arm using basic descriptive statistics.
Readmission due to Wound Complications | Within 30 days of cesarean delivery/wound dressing application
  Hospital readmission events occurring within 30 days postoperatively that are attributable to wound-related issues, including surgical site infection or wound breakdown will be summarized by study arm using basic descriptive statistics.
Reoperation due to Wound Complications | Within 30 days of cesarean delivery/wound dressing application
  The occurrence of a return to the operating room for a wound-related complication (e.g., infection, dehiscence, hematoma evacuation) within the 30-day postoperative period, as documented in the medical record, will be summarized by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Doulaveris, Principal Investigator — Montefiore Medical Center
Locations (1):
- Jack D. Weiler Hospital (Einstein Campus), The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) to be shared will include all data that underlie the results reported in any publication arising from the trial. This includes demographic and clinical characteristics, intraoperative details, incidence of surgical site infections and other wound complications, and patient-reported outcomes from the wound dressing satisfaction questionnaire. No personal identifiers will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available beginning 6 months after publication of the primary results and will remain available for 5 years thereafter.
Access Criteria: Qualified researchers affiliated with academic or healthcare institutions may request access to de-identified individual participant data (IPD) and supporting documentation for purposes of secondary analysis or meta-analysis. Requests must include a brief research proposal outlining study aims, methodology, and intended use of the data. Proposals will be reviewed by the study principal investigator and institutional research committee for scientific merit, ethical compliance, and consistency with the informed consent provided to participants. Approved users must sign a data use agreement. Requests and documentation can be submitted via email to the study PI or designated contact at Montefiore Medical Center.

REFERENCES:
- [Background] Talbot GT, Maxwell RA, Griffiths KM, Polenakovik HM, Galloway ML, Yaklic JL. A Risk-Stratified Peri-Operative Protocol for Reducing Surgical Site Infection after Cesarean Delivery. Surg Infect (Larchmt). 2021 May;22(4):409-414. doi: 10.1089/sur.2019.354. Epub 2020 Aug 12. PMID 32783694
- [Background] Davies P, McCarty S, Hamberg K. Silver-containing foam dressings with Safetac: a review of the scientific and clinical data. J Wound Care. 2017 Jun 1;26(Sup6a):S1-S32. doi: 10.12968/jowc.2017.26.Sup6a.S1. PMID 28594320
- [Background] Saijo Y, Cho H, Mitsuwa H, Ogawa R. Multilayered Silver-containing Polyurethane-foam (Mepilex Ag) for Tie-over Bolster Fixation of a Skin Graft. Plast Reconstr Surg Glob Open. 2024 Aug 1;12(8):e6018. doi: 10.1097/GOX.0000000000006018. eCollection 2024 Aug. PMID 39534070
- [Background] Kuo CY, Wootten CT, Tylor DA, Werkhaven JA, Huffman KF, Goudy SL. Prevention of pressure ulcers after pediatric tracheotomy using a Mepilex Ag dressing. Laryngoscope. 2013 Dec;123(12):3201-5. doi: 10.1002/lary.24094. Epub 2013 Jul 29. PMID 23897691
- [Background] Ball TC, Toy KA, Seoighe DS. The Mepilex Ag glove: A novel burn dressing for hands. Burns. 2025 Mar;51(2):107354. doi: 10.1016/j.burns.2024.107354. Epub 2024 Dec 13. No abstract available. PMID 39721240
- [Background] Lisiecki JL, Buta MR, Taylor S, Tait M, Farina N, Levin J, Schulz J, Sangji N, Friedstat J, Hemmila MR, Wang S, Levi B, Goverman J. Efficacy of Mepliex(R) Ag Versus Xeroform(R) As A Split-Thickness Skin Graft Donor Site Dressing: Bad Habits Die Hard. Ann Burns Fire Disasters. 2023 Sep 30;36(3):243-250. eCollection 2023 Sep. PMID 38680433